CLINICAL TRIAL: NCT05656807
Title: My Weight-their Weight: eHealth Intervention for Managing Obesity in Child Care Settings
Brief Title: Evaluation of Child Care Staff Weight Management Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-0257; R01DK128174 (NIH)
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: child care centers; child care provider health; nutrition; physical activity; body weight; behavior change
MeSH Terms: conditions — Obesity; Motor Activity; Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Go NAPSACC (Active Comparator): Centers randomized to Go NAPSACC will receive the traditional Go NAPSACC program. This will include the center director leading the Go NAPSACC effort with support from a Go NAPSACC Implementation advisor. The advisor will orient each center to Go NAPSACC and its online tools and check in monthly with directors as they work through 2 cycles of Go NAPSACC over 6 months. Centers will take self-assessments on nutrition and physical activity, choose 6 goals (3 from each), create action plans, and take action to achieve their chosen goals.
  Interventions: Behavioral: Go NAPSACC
- Go NAPSACC Enhanced (Experimental): Centers randomized to Go NAPSACC Enhanced will receive the traditional Go NAPSACC program as described in the Active Comparator arm. Additionally, child care providers will simultaneously receive a weight management program, Go NAPSACC Cares over 6 months. The health educator will orient providers with the website and its tools and resources. Providers will take a self-assessment and choose a goal of weight maintenance or weight loss. They will go through 18 lessons with accompanying resources. Within the website they will self-monitor their weight, physical activity, and red foods (diet quality). Providers will receive daily tips, weekly reminders via text message or email, and tailored weekly feedback based on their weight management goals and progress.
  Interventions: Behavioral: Go NAPSACC Enhanced

INTERVENTIONS:
Behavioral: Go NAPSACC Enhanced — Centers will receive the Go NAPSACC program as well as an online weight management intervention that focuses on personal weight management strategies. Participants will have access to materials that will support their adoption of evidence-based strategies for their weight management or loss goal. Behavior change strategies used are meant to increase intervention adherence and improve weight loss.
  Other Names: Go NAPSACC Cares
  Arms: Go NAPSACC Enhanced
Behavioral: Go NAPSACC — Go NAPSACC is an online evidence-based behavioral intervention that supports centers as they adopt center-wide healthy weight practices. It anticipates producing change in the child care environment through fostering best practices in center provisions, practices, policies, and professional development around child nutrition and physical activity and in turn foster healthier habits in the children in their care.
  Arms: Go NAPSACC

SUMMARY:
The goal of this 12-month cluster clinical trial is to evaluate if improving child care providers' health behaviors using an online provider weight management program elicits meaningful change in dietary and physical activity behaviors in 2-5-year-old preschool children in their care and the child care environment.

The study sample will include 84 child care centers. Including: 84 center directors, 168 2-5-year-old classroom teachers, 672 2-5-year old children.

Some centers will do only the online Nutrition and Physical Activity Self-Assessment for Child Care (Go NAPSACC) program. This program works with child care center directors to make changes to their center around child nutrition and physical activity to foster healthier habits for the children enrolled in their care. Other centers will do Go NAPSACC Enhanced. This will include center directors doing Go NAPSACC and 2-5 year old teachers doing an online weight management program with support.

Researchers will compare centers in Go NAPSACC with centers in Go NAPSACC Enhanced to see if there are greater improvements in children's diet quality and physical activity, as well as the nutrition and physical activity environment of centers in the Go NAPSACC Enhanced group. Additionally, they will see if there are greater improvements in teachers' weight, diet quality, and physical activity in centers using Go NAPSACC Enhanced.

DETAILED DESCRIPTION:
This study is a two-group clustered randomized trial to evaluate if improving child care providers' health behaviors elicit meaningful change in dietary and physical activity behaviors in 2-5-year-old preschool children in their care and the child care environment. The investigators will randomize (by center, 1:1 ratio) 84 child care centers, 168 child care providers, and 672 children from these centers to one of two groups (standard Go NAPSACC or Go NAPSACC enhanced) for a 12 month trial (6 months provider weight loss; 6 months no contact follow-up). The specific aims are to 1) improve dietary quality and physical activity behaviors of 2-5-year-old children. 2) improve weight and weight related behaviors (dietary intake and physical activity) of child care providers, and 3) improve the nutrition and physical activity environments at child care centers. Participants randomized to standard Go NAPSACC will receive support for center wide changes focusing on engaging center directors and orienting them to Go NAPSACC, given access to interactive online tools that guide change, and providing ongoing support as they work to adopt evidence-based healthy weight practices. Participants randomized to Go NAPSACC enhanced will receive the traditional Go NAPSACC program (previously described); in addition, child care providers will receive a weight management intervention. The weight management intervention will be guided by social cognitive theory and integrate techniques known to be most effective for changing diet and physical activity behaviors, including intention formation, goal setting (≥5% weight loss at 6 mos. and no regain at 12 mos.), self-monitoring (diet, physical activity, weight), and feedback. Participants will receive a progressive physical activity program. The physical activity program (walking, jogging, biking, etc.) will be progressive and prescribed at a moderate intensity as recommended the "Physical Activity Guidelines for Americans" of 150 min/wk. Starting active minutes goal will be based on self-reported current activity levels: 0 min/wk = 10 min/day goal; 1-59 min/wk = 15/min/day goal, >60 min/wk = 20 min/day goal. The reduced energy diet will follow the Stop Light Diet approach which categorizes foods by energy content: green (low energy: consume freely), yellow (moderate energy: consume in moderation) and red (high energy: consume sparingly). Starting weight will be used to suggest tailored red food limits: Weight Loss - <250lbs = 3; 250 - <300 = 4; >300 = 5. Weight Maintenance - <250 = 4; 250 - <300 = 5; >300 = 6. The stop light diet approach is suitable for all participants (including for whom weight loss may not be recommended [e.g., BMI <25 kg/m2] as it does not specifically prescribe a calorie deficit but focuses on improvement of diet quality.The effectiveness of the intervention will be evaluated by comparing differences between the Go NAPSACC enhanced and standard Go NAPSACC control groups in child's physical activity and diet quality at 6 mos. (primary outcomes). Primary and secondary aims will be analyzed using maximum likelihood methods. Multi-level linear mixed models with repeated measures will be used to estimate change at 6 and 12 mos. and to test for statistical differences across groups in changes over time. Models will include random effect for cluster to account for covariance between participants within the same center as well as fixed effects for time, trial arm, time*arm interaction. To further explore the effect of the intervention, these analyses will be followed by sensitivity analyses that adjust for baseline variables distributed differently between intervention groups and examine completers only. Secondary outcomes will also be examined as longitudinal covariates and asses their association with longitudinal measures of primary outcomes, controlling for treatment, at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Child Care Centers:

* Be open year-round
* Licensed with no plans to close in the next 2 years
* Been in operation for at least 1 year
* Have at least two classrooms serving children 2-5 years-old
* Serve at least lunch to the 2-5-year old children
* Have no history of Go NAPSACC participation in the past 6 months
* Two 2-5-year-old classroom providers and 4 parents from each classroom must provide consent to participate in the study

Child Care Providers (Directors and Teachers):

* Ability to provide informed consent.
* Age 18 years or older.
* Teacher only: Be a teacher in a 2-5-year-old classroom.
* Teacher only: Not pregnant, nor planning to become pregnant in the next year

Children:

* Be in a classroom with a participating child care teacher.
* Be 2-5 years old.
* The consenting primary caregiver must be able to read English

Exclusion Criteria:

Child Care Centers:

* Serve only non-English speaking families

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Diet Quality at Child Care from Baseline to 6 months | Baseline and 6 months post-intervention
  Dietary intake of food consumed by 2-5-year-old children will be assessed via the Diet Observation in Child Care (DOCC) by a trained and certified data collector in the 2-5-year old classroom. Dietary intake data will be used to calculate Healthy Eating Index 2015 (HEI2015) scores to produce an estimate of children's diet quality. Scores range from 0-100, where scores closer to 100 indicate higher diet quality.
Change in Children's Non-sedentary Time at Child Care from Baseline to 6 months | Baseline and 6 months post-intervention
  Physical activity of children 2-5-years old will be assessed by a GT3X+ accelerometer. Children are fitted on the first day of data collection and wear the accelerometer on their non-dominant wrist for 24 hours per day over 7 consecutive days. Cut-points developed for preschool-aged children will be applied to children's accelerometer data to calculate minutes spent in different levels of physical activity (total non-sedentary, sedentary, light, moderate, and vigorous). Non-sedentary time (light, moderate, and vigorous combined) is the primary outcome for this study.

SECONDARY OUTCOMES:
Change in Children's Diet Quality at Child Care from 6 to 12 months | 6 months post-intervention and 12 months post-intervention
  Dietary intake of food consumed by 2-5-year-old children will be assessed via the Diet Observation in Child Care (DOCC) by a trained and certified data collector in the 2-5-year old classroom. Dietary intake data will be used to calculate Healthy Eating Index 2015 (HEI2015) scores to produce an estimate of children's diet quality. Scores range from 0-100, where scores closer to 100 indicate higher diet quality.
Change in Children's Non-sedentary Time at Child Care from 6 to 12 Months | 6 months post-intervention and 12 months post-intervention
  Physical activity of children 2-5-years old will be assessed by a GT3X+ accelerometer. Children are fitted on the first day of data collection and wear the accelerometer on their non-dominant wrist for 24 hours per day over 7 consecutive days. Cut-points developed for preschool-aged children will be applied to children's accelerometer data to calculate minutes spent in different levels of physical activity (total non-sedentary, sedentary, light, moderate, and vigorous). Non-sedentary time (light, moderate, and vigorous combined) is the physical activity outcome.
Change in Child Care Providers Diet Quality | Baseline through 12 months post intervention
  Dietary intake of food consumed by child care providers will be assessed by self-report through the Automated Self-Administered Dietary Assessment Tool (ASA24) over 2 weekdays and 1 weekend day. Dietary intake data will be used to calculate Healthy Eating Index 2015 (HEI2015) scores to produce an estimate of children's diet quality. Scores range from 0-100, where scores closer to 100 indicate higher diet quality. Assessed at baseline and post-intervention at months 6 and 12.
Change in Child Care Providers Physical Activity | Baseline through 12 months post intervention
  Physical activity of child care providers will be assessed by a GT3X+ accelerometer. Child care providers are fitted on the first day of data collection and wear the accelerometer on their non-dominant wrist for 24 hours per day over 7 consecutive days. Cut-points developed for adults will be applied to child care providers accelerometer data to calculate minutes spent in different levels of physical activity (sedentary, light, moderate, and vigorous). Assessed at baseline and post-intervention at months 6 and 12.
Change in Child Care Providers weight | Baseline through 12 months post intervention
  Anthropometrics will be collected in the morning of the onsite visit while participants are in light clothing with shoes removed. Weight will be measured to the nearest 0.1 kg using a Seca digital scale (calibrated quarterly; seca, Chino, CA). Assessed at baseline and post-intervention at months 6 and 12.
Change in Nutrition Environment Score | Baseline through 12 months post intervention
  Each center's nutrition environment will be assessed by trained and certified data collectors who spend two days at the center in a participating classroom using the Environment and Policy Assessment and Observation (EPAO) and Document Review. An overall nutrition environment score will be derived with scores ranging from 0-21, where higher scores indicate better (more supportive) nutrition and physical activity environments. Assessed at baseline and post-intervention at months 6 and 12.
Change in Physical Activity Environment Score | Baseline through 12 months post intervention
  Each center's physical environment will be assessed by trained and certified data collectors who spend two days at the center in a participating classroom using the Environment and Policy Assessment and Observation (EPAO) and Document Review. An overall physical activity environment score will be derived with scores ranging from 0-36, where higher scores indicate better (more supportive) nutrition and physical activity environments. Assessed at baseline and post-intervention at months 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Willis, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center for Health Promotion and Disease Prevention, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina-Chapel Hill (UNC-CH).
Time Frame: Beginning at 9 months and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC-CH.

REFERENCES:
- [Derived] Willis EA, Burney R, Hales D, Ilugbusi LO, Tate DF, Nezami B, Clarke EC, Moore RH, Mathews E, Thompson M, Beckelheimer B, Ward DS. "My wellbeing-their wellbeing "- An eHealth intervention for managing obesity in early care and education: Protocol for the Go NAPSACC Cares cluster randomized control trial. PLoS One. 2023 Jul 7;18(7):e0286912. doi: 10.1371/journal.pone.0286912. eCollection 2023. PMID 37418363